CLINICAL TRIAL: NCT04013906
Title: Randomized Comparison of Rotational Atherectomy vs INtravascular Lithotripsy for Plaque Modification Before Stent implantatiOn in Patients With Severely Calcified Coronary Lesions: The RAINBOW Trial
Brief Title: Atherectomy vs Intravascular Lithotripsy
Acronym: RAINBOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/D/389
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; calcium; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotational atherectomy (Experimental): Patients will undergo rotational atherectomy
  Interventions: Diagnostic Test: Rotational atherectomy
- Intravascular lithotripsy (Experimental): Patients will undergo intravascular lithotripsy
  Interventions: Diagnostic Test: Rotational atherectomy

INTERVENTIONS:
Diagnostic Test: Rotational atherectomy — Rotational atherectomy

SUMMARY:
Preliminary experiences show that IVL is promising for achieving an effective plaque modification at time of PCI.

However, uncertainty about the optimal tool to select in case of calcification of coronary lesions exists, as no randomized comparisons between rotational atherectomy and intravascular lithotripsy have been carried out so far.

The aim of this pilot randomized trial is to evaluate the efficacy and safety of intensive plaque modification with rotational atherectomy vs. intravascular lithotripsy before placement of a drug-eluting stent.

DETAILED DESCRIPTION:
Calcification of the coronary lesion is challenging during percutaneous coronary intervention (PCI) since it can cause the balloon dilation to fail with subsequent incomplete and asymmetrical stent expansion. Also, calcified coronary lesions are associated with increased risk of adverse events after PCI, such as stent restenosis and thrombosis.

Several devices and techniques have been proposed to treat severely calcified coronary lesions. For many years, modification of these lesions with rotational atherectomy has been considered the gold standard to ease the process of angioplasty and PCI. Recently, intravascular lithotripsy (IVL) has been proposed as an alternative to rotational atherectomy for the treatment of calcified de-novo coronary lesions. The Shockwave Medical Coronary Rx Intravascular Lithotripsy (IVL) System (Shockwave Medical Inc., Fremont, California, USA) is a novel balloon catheter-based device able to disrupt calcified lesions using technology like lithotripsy for kidney stones. Preliminary experiences show that IVL is promising for achieving an effective plaque modification at time of PCI.

However, uncertainty about the optimal tool to select in case of calcification of coronary lesions exists, as no randomized comparisons between rotational atherectomy and intravascular lithotripsy have been carried out so far.

The aim of this pilot randomized trial is to evaluate the efficacy and safety of intensive plaque modification with rotational atherectomy vs. intravascular lithotripsy before placement of a drug-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* Reference vessel diameter of 2.5-4.0 mm and lesion lengths of 40 mm or less involving a de novo coronary stenosis.
* Vessel calcification must be severe angiographically as evidenced by calcium present on both sides of the vessel and extending ≥15 mm or by Intravascular ultrasound (IVUS) or optical coherence tomography (OCT) with presence of a calcium arc ≥270° in at least one cross-section.
* Calcifications should not be unable to cross with a balloon

Exclusion Criteria:

• Patients with acute coronary syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | Up to 30 days
  The time to first occurrence of cardiovascular death, non-fatal myocardial infarction, ischemic stroke or ischemia-driven revascularization

SECONDARY OUTCOMES:
Optical coherence tomography (OCT) | Up to 1 day
  The acute lumen gain as assessed by OCT in the two groups

IPD SHARING:
Plan to Share IPD: Undecided